CLINICAL TRIAL: NCT01918878
Title: A 7-month, Multicenter Study to Evaluate the Efficacy of Intravitreal Injections of Aflibercept (EYLEA) 2mg /0.05 ml as Secondary or Third Line Treatment for Neovascular Age-related Macular Degeneration (NVAMD).
Brief Title: Aflibercept (EYLEA)as Secondary or Third Line Treatment for Neovascular Age-related Macular Degeneration.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHO123-HMO-CTIL
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-09

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: age-related macular degeneration; intravitreal injections; Aflibercept; EYLEA
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (EYLEA) (Experimental): Intravitreal injection of aflibercept (EYLEA) 2mg/0.05ml at enrolment (day 0), 4 weeks, 8 weeks, 16 weeks and 24 weeks. Aflibercept will be provided for total period of 24 weeks
  Interventions: Drug: Aflibercept (EYLEA)

INTERVENTIONS:
Drug: Aflibercept (EYLEA) — INTARAVITREAL INJECTION OF AFLIBERCEPT
  Other Names: EYLEA

SUMMARY:
This is a prospective, multicenter, single arm study. The study group will be compose of NVAMD patients who had partial or complete failure responding to initial bevacizumab or ranibizumab treatment of 3-6 monthly intravitreal injections. The patients in the study groups will receive 5 intravitreal injections of aflibercept 2mg/0.05ml at specific visits. Aflibercept will be provided for total period of 24 weeks.

DETAILED DESCRIPTION:
The aim of this study is to prospectively evaluate the use of aflibercept in patients in whom initial incomplete response or loss of initial response for other intravitreal anti- vascular endothelial growth factor (anti-VEGF) therapy was demonstrated.

This is a multi-center study initiated and conducted by the Israeli retina association. Each center participating in the study will follow the same protocol including standardized measurement of visual acuity, OCT, and Fluorescein angiography (FA).

We will enroll 48 NVAMD patients which are partial or non-responded for 3-6 injections of intravitreal bevacizumab or ranibizumab and no more than one year of treatment .

Test Treatment:

Monthly intravitreal aflibercept 2mg /0.05 ml will be given at enrolment (day 0), 4 weeks, 8 weeks, 16 weeks, and 24 weeks after the initial enrollment for the study group.

Follow-up period will be 28 weeks,7 visits. At the 28 week visit the primary and secondary end points will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Ophthalmic Inclusion Criteria

1. Failure of previous intravitreal bevacizumab or ranibizumab treatment, defined as:

   * 3-6 intravitreal injections (The last 3 injections must be no more than 6 weeks between one injection to another).
   * Maximal central thickness by Heidelberg OCT has to be at least 300 microns or larger (retinal thickness including subretinal fluid {SRF},intraretinal fluid {IRF} and PED).
2. Subfoveal choroidal neovascularization (CNV) due to AMD as documented by fluorescein angiogram.
3. Best corrected visual acuity in the study eye between 20/40 and 20/360, inclusive. The VA must be re-confirmed at Day 0 prior to initiation of treatment.
4. Total area of the lesion (including blood, neovascularization, and scar/atrophy) must be ≤ 5 disc areas (DA), of which at least 50% must be active CNV. Active CNV is defined as the neovascular component of the lesion as defined by the fluorescein angiogram.
5. Presence on OCT of subretinal, intraretinal or sub-retinal pigment epithelial (RPE) fluid and/or subretinal thickening consistent with active CNV.
6. Clear ocular media and adequate pupillary dilatation
7. Intraocular pressure (IOP) of 21 mmHg or less.

General Inclusion Criteria

1. Subjects of either gender, aged above 50 years.
2. Women should be post-menopausal for at least 12 months prior to trial entry, or surgically sterile.
3. Provide written informed consent.
4. Ability to comply with study and follow-up procedures and return for all trial visits.

   -

Exclusion Criteria:

Ophthalmic Exclusion Criteria

1. More than 50% of the total lesion size consisting of subretinal hemorrhage.
2. Presence of retinal angiomatous proliferation (RAP).
3. Presence of pigment epithelial tears.
4. Hypersensitivity to the active substance aflibercept or to any of the excipients.
5. Active or suspected ocular or periocular infection.
6. Active severe intraocular inflammation (≥ trace cell or flare), significant epiretinal membrane or vitreomacular traction, macular hole or vitreous hemorrhage.
7. Aphakia or absence of the posterior capsule. Absence of an intact posterior capsule is allowed if it occurred as a result of YAG laser posterior capsulotomy in association with prior posterior chamber intraocular lens (IOL) implantation.
8. History of idiopathic or autoimmune-associated uveitis in either eye.
9. Significant media opacities, including cataract, which might interfere with visual acuity, assessment of toxicity, or fundus photography in the study eye. Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 7 months.
10. Presence of other causes of choroidal neovascularization, including pathologic myopia (spherical equivalent of -8 diopters or more), the ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis.
11. Any intraocular surgery or thermal laser within three (3) months of trial entry.
12. History of any of the following conditions or procedures in the study eye: rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant.
13. Previous therapeutic radiation in the region of the study eye.

General Exclusion Criteria

1. Any of the following underlying diseases including:

1. Clinically significant impaired renal (serum creatinine >2.5 mg/dl or s/p renal transplant or receiving dialysis) or hepatic function.
2. Stroke (within 3 months of trial entry).
3. Any major surgical procedure within one month of trial entry.

2. Any treatment with an investigational agent in the 60 days prior to trial entry for any condition.

3. Known serious allergies to the fluorescein dye used in angiography (mild allergy amenable to treatment is allowable), to the components of the bevacizumab, or aflibercept formulation.

4. Women of child-bearing potential.

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness change | at week 28
  Central macular thickness change from baseline on optical coherence tomography (OCT) at week 28.

SECONDARY OUTCOMES:
change in best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity and Change in CNV size | at week 28
  1. The mean change in best corrected ETDRS visual acuity at 4 meters according to a standardized protocol.
  2. Gain or loss of 3-lines of visual acuity as defined above.
  3. Change in CNV size according to fluorescein angiogram, following a standardized protocol.

OTHER OUTCOMES:
Presence or intraretinal fluid, sub-retinal fluid, or pigment epithelial detachment . | at week 28

CONTACTS AND LOCATIONS:
Overall Officials: Itay Chowers, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel